CLINICAL TRIAL: NCT05772091
Title: Valeur Pronostique Dans Une Population d'Amylose Cardiaque Des paramètres échocardiographiques basée Sur Une Approche d'Apprentissage Automatique
Brief Title: Prognostic Value of Echocardiographic Parameters Based on Machine Learning Approach
Acronym: ATTR-AI
Status: Recruiting | Type: Observational
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2022PI171
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Transthyretin Cardiac Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transthyretin cardiac amyloidosis is an increasingly recognized cause of heart failure with preserved ejection fraction. Its diagnosis is currently based on a non-invasive method including biology and imaging. Still currently incurable, the evolution of this pathology is burdened by numerous comorbidities, including iterative hospitalizations for heart failure leading to death. The Machine Learning approach has already shown its efficiency in terms of diagnosis but its prognostic approach has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of transthyretin cardiac amyloidosis
* Age ≥18 years

Exclusion Criteria:

* Lack of data to confirm or overturn the transthyretin amyloidosis diagnostic
* Echocardiographic data not allowing deep analysis (technical default, bad echogenicity of the patient)
* Final diagnostic of AL or AA amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were managed at participating centers for suspected cardiac amyloidosis or patients with suspected cardiac amyloidosis during hospitalization for another cause.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of death from all causes | Minimum 1-year follow-up and until last news available
  composite endpoint: rate of death from all causes and hospitalisation for acute heart failure following inclusion (with outcome 2
Rate of hospitalisation for acute heart failure | Minimum 1-year follow-up and until last news available
  composite endpoint: rate of death from all causes and hospitalisation for acute heart failure following inclusion (with outcome 1)

SECONDARY OUTCOMES:
Rate of death from all causes | Minimum 1-year follow-up and until last news available
Rate of hospitalisation for acute heart failure (including repeated hospitalisation) | Minimum 1-year follow-up and until last news available
Implantation of pacemaker/defibrillator during study | Minimum 1-year follow-up and until last news available
Rate of death from all causes and hospitalisation for acute heart failure | Minimum 1-year follow-up and until last news available
  composite endpoint: Rate of death from all causes and hospitalisation for acute heart failure, rate of death from all causes and rate of hospitalisation for acute heart failure following inclusion (with outcome 7 and )
Rate of death from all causes | Minimum 1-year follow-up and until last news available
  composite endpoint: Rate of death from all causes and hospitalisation for acute heart failure, rate of death from all causes and rate of hospitalisation for acute heart failure following inclusion (with outcome 6 and 8)
Rate of hospitalisation for acute heart failure | Minimum 1-year follow-up and until last news available
  composite endpoint: Rate of death from all causes and hospitalisation for acute heart failure, rate of death from all causes and rate of hospitalisation for acute heart failure following inclusion (with outcome 6 and 7)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD, PhD, Study Chair — CHRU of Nancy
Locations (4):
- France (4):
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - CHRU de Nancy, Nancy
  - CHU de Rennes Hôpital Pontchaillou, Rennes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No